CLINICAL TRIAL: NCT02759614
Title: Randomized, Open-label, Controlled Multicenter Study to Compare Bevacizumab in Combination With Erlotinib Versus Erlotinib Alone in Chinese NSCLC Patients Harbouring Activating EGFR Mutations(Artemis)
Brief Title: Compare Bevacizumab in Combination With Erlotinib Versus Erlotinib Alone in NSCLC Patients Activating EGFR Mutations
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG1509
Record Dates: First submitted 2016-03-11; First posted 2016-05-03 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: NSCLC
MeSH Terms: interventions — Bevacizumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bevacizumab and Erlotinib (Experimental): Bevacizumab 15 mg/kg shall be intravenous infusion on day 1 once every 3 weeks, Erlotinib 150 mg tablets shall be administered orally every day at least one hour before or two hours after the ingestion of food.
  Interventions: Drug: Bevacizumab; Drug: Erlotinib
- Erlotinib (Active Comparator): Erlotinib 150 mg tablets shall be administered orally every day at least one hour before or two hours after the ingestion of food.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab15mg/kg by intravenous drip infusion on day 1 of a 21-day (within 3 days) cycle and Erlotinib orally once daily at 150mg/day
  Other Names: Avastin
  Arms: Bevacizumab and Erlotinib
Drug: Erlotinib — Erlotinib 150mg, orally once a day
  Other Names: Tarceva

SUMMARY:
This is a randomized, open-label, controlled, multicenter, Phase III study. Patients will be randomly assigned to treatment group (1:1) through a dynamic randomization process with use of the following stratification factors: sex (female/male), disease stage (stage IIIb vs. stage IV vs. recurrence), and EGFR gene mutation (exon 19 deletion vs. exon 21 L858R).

DETAILED DESCRIPTION:
This is a randomized, open-label, controlled, multicenter, Phase III study. Patients will be randomly assigned to treatment group (1:1) through a dynamic randomization process with use of the following stratification factors: sex (female/male), disease stage (stage IIIb vs. stage IV vs. recurrence), and EGFR gene mutation (exon 19 deletion vs. exon 21 L858R).

An independent review committee (IRC) will be used to determine the response based study endpoints. IRC membership and procedures will be detailed in an IRC charter.

A data safety monitoring board (DSMB) will be used in this study. DSMB is an independent body and will be responsible for reviewing safety data of the study. DSMB membership and procedures will be detailed in a separate DSMB document.

Information regarding the nature and the duration of subsequent treatment will be collected.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria for study entry:

1. Signed Informed Consent Form.
2. Age≥18 years.
3. Able to comply with the study protocol, in the investigator's judgment.
4. Histologically or cytologically documented inoperable, locally advanced (Stage IIIb who are not amenable for combined modality treatment), metastatic (Stage IV) or recurrent non-squamous NSCLC. Diagnoses of non-squamous NSCLC based on sputum cytology alone are not acceptable.
5. An exon 19 deletion mutation or exon 21 L858R mutation has been found in high-sensitivity EGFR mutation tests by PCR using tumor tissue centrally confirmed. Direct sequencing is not accepted.
6. Eastern Cooperative Oncology Group performance status 0-1.
7. Life expectancy≥12 weeks.
8. Previous systemic cytotoxic chemotherapy for locally advanced, metastatic or recurrent disease has not been performed. Subjects who have undergone intracavity administration with an antineoplastic agent during pleurodesis are not permitted. For patients who have undergone pre- or postoperative adjuvant chemotherapy, at least 6 months have elapsed since the final administration date.
9. Patients who have undergone radiotherapy may be enrolled if they meet the following conditions:

   * The patient has no history of radiotherapy for lesions in lung fields within 28 days before the randomization.
   * For radiotherapy outside the chest region, at least 28 days have elapsed by the time of randomization since the final irradiation date. (if the radiotherapy given as palliation to bone metastases within 2 weeks, the patient should recovery from all toxicities)
10. Measurable disease at baseline. At least one lesion is present that can be measured in accordance with the criteria in Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. However, sites treated by radiotherapy should not be considered measurable.
11. Adequate haematological function:

    * Absolute neutrophil count (ANC)≥1.5×109/L AND
    * Platelet count≥100×109/L AND
    * Haemoglobin≥9 g/dL (may be transfused to maintain or exceed this level)
12. Adequate liver function.

    * Total bilirubin<1.5×upper limit of normal (ULN) AND
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)<2.5×ULN in patients without liver metastases; <5×ULN in patients with liver metastases
13. Adequate renal function

    * Serum creatinine≤1.5×ULN or calculated creatinine clearance≧45mL/min AND
    * Urine dipstick for proteinuria<2+. Patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate≤1 g of protein in 24 hours.
14. International normalised ratio (INR)≤1.5 and partial prothrombin time (PTT or aPTT)≤1.5×ULN within 7 days prior to randomization.
15. For women who are not postmenopausal (≥12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use single or combined contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the last dose of study drug.
16. For men: agreement to remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the last dose of study drug and agreement to refrain from donating sperm during this same period.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

1. Mixed adenosquamous carcinomas with predominantly squamous component.
2. A positive result for the exon 20 T790M mutation from any high-sensitivity EGFR mutation test such as digital PCR using tumor tissue or cells.
3. Evidence of CNS metastases, except for the patients without any symptom or the patients with symptom but have stable disease for at least 28 days after treatment of CNS metastases.
4. History of haemoptysis, defined as > 2.5 ml of red blood per event within 3 months prior to randomization.
5. Evidence of tumour invading major blood vessels on imaging. The investigator or the local radiologist must exclude evidence of tumour that is fully contiguous with, surrounding, or extending into the lumen of a major blood vessel (e.g., pulmonary artery or superior vena cava).
6. Major surgery (including open biopsy) or significant traumatic injury within 28 days prior to randomization or anticipation of the need for major surgery during study treatment.
7. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device are excluded within 7 days prior to initiation of study treatment. Placement of a vascular access device should be at least 2 days prior to initiation of study treatment.
8. Current or recent (within 10 days of first dose of bevacizumab) use of aspirin (325 mg/day) or other nonsteroidal anti-inflammatory agents known to inhibit platelet function.
9. Current or recent (within 10 days of first dose of bevacizumab) use of full-dose oral or parenteral anticoagulants or thrombolytic agent for therapeutic purposes. Prophylactic use of anticoagulants is allowed.
10. History or evidence of inherited bleeding diathesis or coagulopathy that increases the risk of bleeding.
11. Uncontrolled hypertension (blood pressures: systolic>150 mmHg and/or diastolic >100 mmHg).
12. Prior history of hypertensive crisis or hypertensive encephalopathy.
13. Clinically significant (i.e., active) cardiovascular disease, including but not limited to cerebral vascular accident (CVA) or (transient ischemic attack) TIA (≤6 months before randomization), myocardial infarction (≤6 months before randomization), unstable angina, congestive heart failure New York Heart Association Class≥II, or serious cardiac arrhythmia requiring medication during the study and that might interfere with regularity of the study treatment or not controlled by medication.
14. Significant vascular disease (including but not limited to aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to randomization.
15. Non-healing wound, active peptic ulcer, or bone fracture.
16. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months of enrollment.
17. Pregnant or lactating, or intending to become pregnant during the study.
18. Treatment with any other investigational agent or participation in another clinical trial within 28 days prior to randomization.
19. Known hypersensitivity to bevacizumab and Chinese hamster ovary cell products or other recombinant human or humanised antibodies or erlotinib or any of its excipients.
20. Evidence of ongoing or active infection requiring IV antibiotics; any other disease, neurological, or metabolic dysfunction; physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications.
21. Patients diagnosed with a tracheo-oesophageal fistula.
22. Prior chemotherapy or treatment with another systemic anti-cancer agent (e.g., monoclonal antibody, tyrosine kinase inhibitors, EGFR inhibitors, VEGF receptor inhibitors) for the treatment of the patient's current stage of disease (Stage IIIB not amenable for combined modality treatment, Stage IV or postoperative recurrent disease). NOTE:

    i. Previous adjuvant or neo-adjuvant treatment for non-metastatic disease is permitted if completed ≥ 6 months before randomization.
23. Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication, or have active gastroduodenal ulcer disease.
24. Any inflammatory changes of the surface of the eye (e.g.: severe dry eye syndrome, keratoconjunctivitis, keratitis etc.) or any other disorder likely to increase the risk of corneal epithelial lesions. The use of contact lenses is not recommended during the study. The decision to continue to wear contact lenses should be discussed with the patient's treating oncologist and the ophthalmologist.
25. Patients with pre-existing Interstitial Lung Disease or pulmonary fibrosis.
26. Malignancies other than NSCLC within 5 years prior to randomization, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) by IRC | The primary PFS analysis will be performed when approximately 224 PFS events (disease progression or death, whichever occurs first) have occurred, which is estimated to occur at approximately 18 months after enrollment of the last patient.
  To evaluate the efficacy of bevacizumab combined with erlotinib compared with erlotinib alone in patients with NSCLC harbouring activating EGFR mutations, as measured by independent review committee assessed progression-free survival using RECIST v1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) by investigator using RECIST v1.1 | The primary PFS analysis will be performed when approximately 224 PFS events (disease progression or death, whichever occurs first) have occurred, which is estimated to occur at approximately 18 months after enrollment of the last patient.
  To evaluate the efficacy of bevacizumab combined with erlotinib compared with erlotinib alone in patients with NSCLC harbouring activating EGFR mutations, as measured by investigators assessed progression-free survival using RECIST v1.1
Objective response rate (ORR) by IRC using RECIST v1.1 | baseline overall tumor assessment can be performed up to 28 days prior to randomization. Post-baseline assessment will be performed every six weeks until 1st disease progression, through study completion, an average of 2 years.
  To evaluate the efficacy of bevacizumab combined with erlotinib compared with erlotinib alone in patients with NSCLC harbouring activating EGFR mutations, as measured by independent review committee assessed objective response rate using RECIST v1.1
Objective response rate (ORR) by investigator using RECIST v1.1 | baseline overall tumor assessment can be performed up to 28 days prior to randomization. Post-baseline assessment will be performed every six weeks until 1st disease progression, through study completion, an average of 2 years.
  To evaluate the efficacy of bevacizumab combined with erlotinib compared with erlotinib alone in patients with NSCLC harbouring activating EGFR mutations, as measured by investigators assessed objective response rate using RECIST v1.1
Disease control rate (DCR) by IRC using RECIST v1.1 | That is expected to be approximately 57 months.
  Disease control rate (DCR) will be analyzed using similar method as objective response rate.
Disease control rate (DCR) by investigator using RECIST v1.1 | That is expected to be approximately 57 months.
  Disease control rate (DCR) will be analyzed using similar method as objective response rate.
Duration of response(DOR) by IRC using RECIST v1.1 | That is expected to be approximately 57 months.
  Duration of response(DOR) will be analyzed using similar method as objective response rate.
Duration of response(DOR) by investigator using RECIST v1.1 | That is expected to be approximately 57 months.
  Duration of response(DOR) will be analyzed using similar method as objective response rate.
Overall survival(OS) | That is expected to be approximately 57 months.
  To evaluate the efficacy of bevacizumab combined with erlotinib compared with erlotinib alone in patients with NSCLC harbouring activating EGFR mutations, as measured by investigators assessed overall survival .

CONTACTS AND LOCATIONS:
Overall Officials: Qing Zhou, PhD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Lung Cancer Institute, Guangdong General Hospital, Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
DSMB

REFERENCES:
- [Result] Sequist LV, Yang JC, Yamamoto N, O'Byrne K, Hirsh V, Mok T, Geater SL, Orlov S, Tsai CM, Boyer M, Su WC, Bennouna J, Kato T, Gorbunova V, Lee KH, Shah R, Massey D, Zazulina V, Shahidi M, Schuler M. Phase III study of afatinib or cisplatin plus pemetrexed in patients with metastatic lung adenocarcinoma with EGFR mutations. J Clin Oncol. 2013 Sep 20;31(27):3327-34. doi: 10.1200/JCO.2012.44.2806. Epub 2013 Jul 1. PMID 23816960
- [Result] Seto T, Kato T, Nishio M, Goto K, Atagi S, Hosomi Y, Yamamoto N, Hida T, Maemondo M, Nakagawa K, Nagase S, Okamoto I, Yamanaka T, Tajima K, Harada R, Fukuoka M, Yamamoto N. Erlotinib alone or with bevacizumab as first-line therapy in patients with advanced non-squamous non-small-cell lung cancer harbouring EGFR mutations (JO25567): an open-label, randomised, multicentre, phase 2 study. Lancet Oncol. 2014 Oct;15(11):1236-44. doi: 10.1016/S1470-2045(14)70381-X. Epub 2014 Aug 27. PMID 25175099
- [Result] Maemondo M, Inoue A, Kobayashi K, Sugawara S, Oizumi S, Isobe H, Gemma A, Harada M, Yoshizawa H, Kinoshita I, Fujita Y, Okinaga S, Hirano H, Yoshimori K, Harada T, Ogura T, Ando M, Miyazawa H, Tanaka T, Saijo Y, Hagiwara K, Morita S, Nukiwa T; North-East Japan Study Group. Gefitinib or chemotherapy for non-small-cell lung cancer with mutated EGFR. N Engl J Med. 2010 Jun 24;362(25):2380-8. doi: 10.1056/NEJMoa0909530. PMID 20573926